CLINICAL TRIAL: NCT07157215
Title: An International Survey on the Use of NIV Outside the ICU (NIV-Safety Study)
Brief Title: An International Survey on the Use of NIV Outside the ICU
Acronym: NIV-SAFETY
Status: Recruiting | Type: Observational
Sponsor: Dr. Ram Manohar Lohia Hospital (Other Government)
Collaborators: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government); Hamad Medical Corporation (Industry); Instituto Murciano de Investigación Biosanitaria (IMIB) (Unknown)
Responsible Party: Principal Investigator, Sanjay Singhal, sanjay, Dr. Ram Manohar Lohia Hospital
Other Study IDs: RC-2029/RMLIMS/2025/18.08.2025
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Non-invasive Ventilation; Intensive Care (ICU); Safety
Keywords: NIV; SAFETY; ICU

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PROFESSIONAL USING NIV: physicians, nursing officers, and Respiratory therapists who treat patients with NIV

SUMMARY:
Non-invasive ventilation (NIV) is a way to support breathing using a mask or helmet instead of a breathing tube, and it is proven to reduce the need for intubation, save lives, shorten hospital stays, and lower costs. While NIV has long been used in intensive care units, it is now increasingly applied in emergency rooms, hospital wards, and long-term care facilities. However, global data on how it is used outside ICUs-such as which patients receive it, how well it works, and what barriers exist-is lacking. The NIV-Safety Study is a worldwide survey of doctors, nurses, and respiratory therapists to understand current practices, outcomes, and challenges of NIV use beyond the ICU. The findings aim to guide safer, more effective, and standardized use of NIV across different healthcare settings.

DETAILED DESCRIPTION:
BACKGROUND Non-invasive ventilation (NIV) has been an essential tool in respiratory care since its introduction and remains a cornerstone in managing respiratory failure. Evidence-based guidelines recommend NIV as the first-line treatment for acute episodes in four key conditions: COPD exacerbations, cardiogenic pulmonary edema, pulmonary infiltrates in immunocompromised patients, and as a weaning strategy for COPD patients post-extubation [1]. Over the years, NIV has been widely adopted for managing acute respiratory failure across various conditions [2]. It is an effective alternative to invasive mechanical ventilation, helping to prevent intubation and reducing the risk of reintubation after extubation. While traditionally used in intensive care units (ICUs), its application has expanded beyond the ICU to settings such as emergency departments, general wards, high-dependency units (HDUs), and long-term care facilities [3]. Early initiation of NIV has been shown to reduce the need for intubation, lower mortality rates in acute COPD exacerbations, and decrease both hospital costs and length of stay [4]. Despite these benefits, several challenges persist, including inconsistencies in clinical protocols, inadequate staff training, and disparities in resource availability across healthcare systems. Additionally, there is a significant gap in comprehensive global data on NIV use and patient outcomes in non-ICU settings [5]. Understanding the international landscape of NIV implementation, including current practices, protocols, and barriers, is essential for optimizing patient care and establishing standardized guidelines. The NIV-Safety Study aims to bridge this gap by evaluating the prevalence of non-invasive ventilation (NIV) use outside the intensive care unit (ICU), global trends, indications, and challenges associated with NIV use outside the ICU.

RATIONALE FOR CURRENT STUDY:

Early initiation of NIV has been shown to reduce the need for intubation, lower mortality rates in acute COPD exacerbations, and decrease both hospital costs and length of stay [4]. While traditionally used in intensive care units (ICUs), its application has expanded beyond the ICU to settings such as emergency departments, general wards, high-dependency units (HDUs), and long-term care facilities [3]. Despite these benefits, several challenges persist, including inconsistencies in clinical protocols, inadequate staff training, and disparities in resource availability across healthcare systems. Additionally, there is a significant gap in comprehensive global data on NIV use and patient outcomes in non-ICU settings [5]. Understanding the international landscape of NIV implementation, including current practices, protocols, and barriers, is essential for optimizing patient care and establishing standardized guidelines. To date, no study has examined the use of NIV outside the ICU. A lack of data hampers the transfer of the benefits of scientific research to patients. This study aimed to evaluate global trends, indications, and challenges associated with NIV use outside the ICU.

OBJECTIVE

1. Primary To assess the prevalence of non-invasive ventilation (NIV) use outside the ICU
2. Secondary

   1. To identify the common conditions treated with NIV in non-ICU settings.
   2. To evaluate the outcomes of using NIV in non-ICU settings.
   3. To examine the barriers and challenges healthcare providers face when using NIV outside the ICU.

METHODOLOGY

1. Study design This cross-sectional, multi-national, web-based survey of physicians, nursing officers, and Respiratory therapists who treat patients with NIV will be conducted after approval from the Institutional Ethics Committee (IEC) of the Dr Ram Manohar Lohia Institute of Medical Sciences, Lucknow. Participation will be on an invitation basis and purely voluntary, after informed consent.
2. Inclusion criteria Physicians, Nursing Officers, and Respiratory therapists dealing with adult patients with acute and chronic respiratory failure.
3. Exclusion Criteria Physicians and Respiratory therapists who refuse to give consent.
4. Study Protocol:

   A pre-designed survey link will be sent to all members of various respiratory and critical care societies, as well as institutions/hospitals. Each physician, nursing officer, and RT who consented to participate will receive a web-based questionnaire. Those who did not respond to the first email within eight weeks will receive reminders.
5. Definitions:

   NIV stands for non-invasive ventilation. It is the application of respiratory support via a sealed face mask, nasal mask, or helmet mask via a portable BIPAP, CPAP, or ICU ventilator.

   A pre-designed survey link (https://forms.gle/6mJyw172MxSVdbxP8) will be sent Wait for 8 weeks If there is no response, a reminder will be sent
6. Outcome measures:

a) prevalence of non-invasive ventilation (NIV) uses outside the intensive care unit b) Data collection: Demographic and clinical characteristics of all eligible patients will be collected on a structured web form.

(https://forms.gle/6mJyw172MxSVdbxP8) g) Sample size and statistical analysis: According to a study by Walkey AJ et al. [6], the proportion of COPD patients who received NIV was 12.3%. We calculated our sample size using the formula N = t²·p·q / ε², where N is the required sample size, t corresponds to the 95% confidence level (standard value of 1.96), p is the estimated prevalence, q is one minus the prevalence, and ε represents the allowable error. Applying this formula with a prevalence of 12.3%, our initial sample size is 166. To enhance validity, we increased the sample size by 20%, resulting in a final sample size of 199. Since we have three groups of responders (Physicians, Nurses, and Respiratory Therapists), we maintained a minimum total sample size of 600. Data will be collected, compiled, and analyzed using IBM SPSS 21 software. Quantitative data will be analyzed by measuring central tendencies, including the mean, standard deviation, standard error, confidence interval, and median. Qualitative data will be analyzed using Fisher's exact test, the Chi-square test (with Yates' correction if needed), and Spearman's rank correlation test.

h) Study duration: 06 months i) Study registration: After IEC approval, this study will be registered at clinicaltrials.gov.in.

j) ETHICAL CONSIDERATION: No intervention is involved in this web-based questionnaire study. Informed Consent will be obtained before the questionnaire is filled out.

k) FINANCIAL ASPECTS: This will be a non-funded observational study. Investigators, collaborators, and patients will not receive incentives or honorarium.

l) Role and Responsibilities: The steering committee will appoint national coordinators (NCs) who will be key in conducting the study in individual countries as project leaders. The role/responsibilities of the NC include the following: Advertise the survey in each country and identify local participants. The PI and Executive Members will use this data solely for scientific purposes. Investigators will be informed about ongoing analyses and related study activities, such as presentations at meetings. All investigators have the right to submit study questions after the analyses described in the protocol have been completed. The Steering Committee will determine whether the proposed analysis can be performed, provided it does not conflict with other ongoing or completed analyses. Data in the database will not be distributed to third parties without the explicit and written agreement of the local investigator.

m) Publication Policy: Steering Committee members and National coordinators will be part of the writing committee and listed as authors of the final manuscript. All local investigators will be kept as collaborators if they have contributed more than 20 responses. Based on patient enrolment, participation in data analysis, and contribution to the final manuscript.

n) REFERENCES

1. Nava S. Behind a mask: tricks, pitfalls, and prejudices for noninvasive ventilation. Respir Care. 2013 Aug;58(8):1367-76. doi: 10.4187/respcare.02457. PMID: 23878302.
2. Vatrella A, Fabozzi I. Non invasive ventilation away from ICU. Transl Med UniSa. 2012 Jan 18;2:64-5. PMID: 23905046; PMCID: PMC3728781.
3. Cabrini L, Idone C, Colombo S, Monti G, Bergonzi PC, Landoni G, Salaris D, Leggieri C, Torri G. Medical emergency team and non-invasive ventilation outside ICU for acute respiratory failure. Intensive Care Med. 2009 Feb;35(2):339-43. doi: 10.1007/s00134-008-1350-y. Epub 2008 Nov 19. PMID: 19018515.
4. Plant PK, Owen JL, Elliott MW. Early use of non-invasive ventilation for acute exacerbations of chronic obstructive pulmonary disease on general respiratory wards: a multicentre randomised controlled trial. Lancet. 2000 Jun 3;355(9219):1931-5. doi: 10.1016/s0140-6736(00)02323-0. PMID: 10859037.
5. Carron M, Freo U, BaHammam AS, Dellweg D, Guarracino F, Cosentini R, Feltracco P, Vianello A, Ori C, Esquinas A. Complications of non-invasive ventilation techniques: a comprehensive qualitative review of randomized trials. Br J Anaesth. 2013 Jun;110(6):896-914. doi: 10.1093/bja/aet070. Epub 2013 Apr 5. PMID: 23562934.
6. Walkey AJ, Wiener RS. Use of noninvasive ventilation in patients with acute respiratory failure, 2000-2009: a population-based study. Ann Am Thorac Soc. 2013 Feb;10(1):10-7. doi: 10.1513/AnnalsATS.201206-034OC. PMID: 23509327; PMCID: PMC3780971.

ELIGIBILITY:
Inclusion criteria Physicians, Nursing Officers, and Respiratory therapists dealing with adult patients with acute and chronic respiratory failure.

Exclusion Criteria Physicians and Respiratory therapists who refuse to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: physicians, nursing officers, and Respiratory therapists who treat patients with NIV
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
prevalence of non-invasive ventilation (NIV) use outside the ICU | SIX MONTHS
  To assess the prevalence of non-invasive ventilation (NIV) use outside the ICU

SECONDARY OUTCOMES:
Common conditions treated with NIV in non-ICU settings | SIX MONTHS
  the common respiratory conditions who are treated with NIV in non-ICU settings.
outcomes of using NIV in non-ICU settings | six months
  Outcome of NIV (success/failure) if used in non-ICU settings
Barriers and challenges faced while using NIV in non-ICU settings | six months
  Barriers and challenges faced by healthcare personals while using NIV in non-ICU settings

OTHER OUTCOMES:
(untitled outcome) | SIX MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, Study Chair — SGPGIMS; Antonio M Esquinas, MD, PhD, FCCP, FNIV, FBCV, Study Chair — Instituto Murciano de Investigacion Biosanitaria,
Locations (1):
- Dr Ram Manohar Lohia Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Access to STUDY IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication of manuscript and the data will be made accessible for up to 24 months
Access Criteria: qualified researchers engaging in independent scientific research

REFERENCES:
- [Background] Walkey AJ, Wiener RS. Use of noninvasive ventilation in patients with acute respiratory failure, 2000-2009: a population-based study. Ann Am Thorac Soc. 2013 Feb;10(1):10-7. doi: 10.1513/AnnalsATS.201206-034OC. PMID 23509327
- [Background] Carron M, Freo U, BaHammam AS, Dellweg D, Guarracino F, Cosentini R, Feltracco P, Vianello A, Ori C, Esquinas A. Complications of non-invasive ventilation techniques: a comprehensive qualitative review of randomized trials. Br J Anaesth. 2013 Jun;110(6):896-914. doi: 10.1093/bja/aet070. Epub 2013 Apr 5. PMID 23562934
- [Background] Plant PK, Owen JL, Elliott MW. Early use of non-invasive ventilation for acute exacerbations of chronic obstructive pulmonary disease on general respiratory wards: a multicentre randomised controlled trial. Lancet. 2000 Jun 3;355(9219):1931-5. doi: 10.1016/s0140-6736(00)02323-0. PMID 10859037
- [Background] Cabrini L, Idone C, Colombo S, Monti G, Bergonzi PC, Landoni G, Salaris D, Leggieri C, Torri G. Medical emergency team and non-invasive ventilation outside ICU for acute respiratory failure. Intensive Care Med. 2009 Feb;35(2):339-43. doi: 10.1007/s00134-008-1350-y. Epub 2008 Nov 19. PMID 19018515
- [Background] Vatrella A, Fabozzi I. Non invasive ventilation away from ICU. Transl Med UniSa. 2012 Jan 18;2:64-5. Print 2012 Jan. No abstract available. PMID 23905046
- [Background] Nava S. Behind a mask: tricks, pitfalls, and prejudices for noninvasive ventilation. Respir Care. 2013 Aug;58(8):1367-76. doi: 10.4187/respcare.02457. PMID 23878302